CLINICAL TRIAL: NCT06554912
Title: Evaluation of Safety and Feasibility of Lymphatic Decompression in Chronic Heart Failure
Brief Title: FLOWS-HF : Feasibility of Lymphatic Offloading with Stenting in Heart Failure
Acronym: FLOW-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: stop financial collaboration
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Selera Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC24.0032
Record Dates: First submitted 2024-04-25; First posted 2024-08-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases; Chronic Heart Failure
Keywords: Lymphatic Decompression; Chronic Heart Failure; Stenting; Lymphatic system
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphatic Decompression (Experimental): Pre-procedural evaluation : CT with contrast injected in the right arm, baseline heart failure questionaries and assessments Study intervention : Transvenous retrograde access of the thoracic duct, hemodynamic measures, measurement of central venous and thoracic duct pressures, lymphovenous junction stenting, fluid sampling Follow-up evaluation : phone calls on days 2 and 7 to assess adverse events and in-person consultations including adverse events, heart failure questionaries and assessments at 1, 3, and 6 months
  Interventions: Procedure: Lymphatic Decompression

INTERVENTIONS:
Procedure: Lymphatic Decompression — Patients will be prepared according to standard procedures Clinical examinations, para-clinical assessment and biological tests Patient will be set in angiography room and local anesthesia at the puncture area (femoral vein or brachial vein).
  Obtain access to the femoral vein per standard procedures (option for brachial access depending on anatomy based on pre-operative CT, per physician discretion) After setting introducer sheath, catheterism of cardiac cavity will be performed for assess the following standard hemodynamic measures Catheterism of thoracic duct through the subclavian vein will be performed under fluoro guidance and phlebography using contrast Measure TD and central venous pressures Deploy stent under fluoro guidance Standard vascular stent deployed in subclavian vein and into lymphovenous junction Evaluate the procedure with standard phlebography and hemodynamic measures Remove catheters, and temporary compression as standard venous procedures

SUMMARY:
The main objective is to evaluate the safety of lymphatic decompression in heart failure.

The research hypothesis is that lymphatic decompression is safe and feasible in heart failure patients with recurrent congestion despite on maximum tolerated diuretic dosage. Safety will be evaluated by the rate and severity of adverse events. Feasibility will be assess based on procedural success and time.

In demonstrating that this approach is both safe and feasible, the expected benefits of the research include symptom relief for patients as well as data generation and considerations for a novel treatment for chronic heart failure patients. Ultimately, this research will contribute to the development of an additional treatment option for patients that remain congested while on standard-of-care therapies.

DETAILED DESCRIPTION:
Better understanding of the lymphatic system's role in managing volume status and how this system is overwhelmed in HF has made it a compelling target for intervention. Historic and contemporary preclinical and clinical evidence demonstrate that surgically relieving or bypassing the resistance at the LVJ when the lymphatic system is overwhelmed significantly improves volume status in heart failure. Although it demonstrates clinical benefit in a majority of patients, the surgical approach has greater risks and is not scalable due to technical difficulties. More recently, improved clinical outcomes and feasibility of minimally invasive lymphatic decompression via transcatheter thoracic duct stenting was demonstrated in cirrhosis, another volume-overload related condition. With supportive preclinical and clinical data, this study aims to evaluate lymphatic decompression in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age
* Diagnosis of chronic heart failure (reduced or preserved EF) with evidence of diastolic dysfunction on echocardiogram
* Chronic NYHA class II or greater
* Prone to cardiorenal syndrome or refractory to diuretics (e.g. on lasix 125 mg PO total daily dose or equivalent diuretic dosing for 1 or more months prior to enrollment)
* History of symptoms of congestion (e.g. dyspnea, peripheral edema, pleural effusion, and/or ascites) in preceding 12 months requiring HF hospitalization with IV diuresis
* NT-proBNP >1000 pg/ml
* eGFR > 20 ml/min/1.73m2
* Life expectancy > 6 months
* Membership of the social security system or benefiting from such a system
* Able and willing to sign informed consent

Exclusion Criteria:

* Anatomy not considered suitable based on CT with contrast (e.g., not visible, multiple terminal ducts or plexiform termination)
* Other cause of thoracic duct congestion based on CT with contrast (superior cava vein/left brachiocephalic vein/ jugular or subclavian vein thrombosis)
* Acute coronary syndrome, stroke, pulmonary embolism in previous 6 months
* Stage IV or stage V chronic kidney disease, or end-stage renal disease (ESRD) requiring dialysis, or severe renal failure (<30ml/min)
* Cardiac surgery within past 6 months (coronary artery bypass grafting, valvular, or pericardial surgery)
* Transcatheter structural heart intervention within past 6 months
* Active pregnancy, breastfeeding, or anticipated pregnancy within 1 year
* Known coagulation disorders or inability to take blood thinning medications (anticoagulation or antiplatelet therapy) for at least one month after procedure
* Severe pulmonary hypertension (RVSP >60mmHg as assessed by echocardiogram)
* Severe RV dysfunction (TAPSE <17mm, RFAC <35%)
* Known allergies or sensitivities to materials utilized in procedure, including contrast agents
* Candidate deemed unsuitable based on investigator opinion
* Subject in exclusion period of another study
* Subject under administrative or judicial supervision
* Subject unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the lymphatic decompression's safety in heart failure by the assessment of the rate and severity of adverse events after the procedure of thoracic duct decompression. | During 180 days after the procedure +/- 4 days
  Assessment of the rate and severity of adverse events after the procedure of thoracic duct decompression.

SECONDARY OUTCOMES:
Evaluation of the lymphatic decompression's feasibility in heart failure | Procedure day (D0-1)
  Lymphatic decompression's success (Y/N)
Evaluation of the lymphatic decompression's feasibility in heart failure | Procedure day (D0-1)
  Procedure time (intervention time in minutes)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (urine output) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including urine output (mL)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (sodium output) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including sodium output (mmol/L/24h)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (medication dosing requirements). | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including medication dosing requirements
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (KCCQ quality of life score) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including KCCQ quality of life score (scaled from 0 to 100 and represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent).
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (EVEREST congestion score) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including EVEREST congestion score (based on specific symptoms and signs ranges from 0 to 3 for each symptom or sign)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (6-min walk test) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including 6-min walk test (The distance in metres walked reflects the patient's functional capacity)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (number of heart failure hospitalization) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including number of HF hospitalization
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (IV diuresis rates) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including IV diuresis rates (mg/day)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (frequency of paracentesis) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including frequency of paracentesis (mg/L)
To evaluate the lymphatic decompression's efficacy in heart failure by change in heart failure symptoms. (frequency of thoracentesis) | During 180 days after the procedure +/- 4 days
  Change in HF symptoms, including frequency of thoracentesis (mg/L)
Evaluation of the lymphatic decompression's impact on thoracic duct pressure | Before the procedure and days 90 +/- 4 days after the procedure
  Change in pressure gradient across lymphovenous junction before and after stenting
Evaluation of the lymphatic decompression's impact on central hemodynamic functions. (Blood flow dynamics in mmHg). | Days 30, Days 90 and days 180 after the procedure
  Changes in hemodynamic measures during intervention evaluated by catheter in right cavities before decompression, 30 minutes after decompression and 3 months after the procedure.
Evaluation of the lymphatic decompression's impact on renal function | Days 30, Days 90 and days 180 after the procedure
  Changes in creatinine / eGFR before and after the procedure (M1, M3, M6).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osenenko KM, Kuti E, Deighton AM, Pimple P, Szabo SM. Burden of hospitalization for heart failure in the United States: a systematic literature review. J Manag Care Spec Pharm. 2022 Feb;28(2):157-167. doi: 10.18553/jmcp.2022.28.2.157. PMID 35098748
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Cotter G, Metra M, Milo-Cotter O, Dittrich HC, Gheorghiade M. Fluid overload in acute heart failure--re-distribution and other mechanisms beyond fluid accumulation. Eur J Heart Fail. 2008 Feb;10(2):165-9. doi: 10.1016/j.ejheart.2008.01.007. PMID 18279771
- [Background] Miller WL. Fluid Volume Overload and Congestion in Heart Failure: Time to Reconsider Pathophysiology and How Volume Is Assessed. Circ Heart Fail. 2016 Aug;9(8):e002922. doi: 10.1161/CIRCHEARTFAILURE.115.002922. PMID 27436837
- [Background] Uduman J. Epidemiology of Cardiorenal Syndrome. Adv Chronic Kidney Dis. 2018 Sep;25(5):391-399. doi: 10.1053/j.ackd.2018.08.009. PMID 30309456
- [Background] Miller WL. Fluid Volume Homeostasis in Heart Failure: A Tale of 2 Circulations. J Am Heart Assoc. 2022 Sep 20;11(18):e026668. doi: 10.1161/JAHA.122.026668. Epub 2022 Sep 8. PMID 36073644
- [Background] Rengstorff RH. Astigmatism after contact lens wear. Am J Optom Physiol Opt. 1977 Nov;54(11):787-91. doi: 10.1097/00006324-197711000-00008. PMID 610440
- [Background] Neuberg GW, Miller AB, O'Connor CM, Belkin RN, Carson PE, Cropp AB, Frid DJ, Nye RG, Pressler ML, Wertheimer JH, Packer M; PRAISE Investigators. Prospective Randomized Amlodipine Survival Evaluation. Diuretic resistance predicts mortality in patients with advanced heart failure. Am Heart J. 2002 Jul;144(1):31-8. doi: 10.1067/mhj.2002.123144. PMID 12094185
- [Background] Shams E, Bonnice S, Mayrovitz HN. Diuretic Resistance Associated With Heart Failure. Cureus. 2022 Jan 18;14(1):e21369. doi: 10.7759/cureus.21369. eCollection 2022 Jan. PMID 35198282
- [Background] Itkin M, Rockson SG, Burkhoff D. Pathophysiology of the Lymphatic System in Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Jul 20;78(3):278-290. doi: 10.1016/j.jacc.2021.05.021. PMID 34266581
- [Background] Fudim M, Salah HM, Sathananthan J, Bernier M, Pabon-Ramos W, Schwartz RS, Rodes-Cabau J, Cote F, Khalifa A, Virani SA, Patel MR. Lymphatic Dysregulation in Patients With Heart Failure: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Jul 6;78(1):66-76. doi: 10.1016/j.jacc.2021.04.090. PMID 34210416
- [Background] Martens P, Tang WHW. Targeting the Lymphatic System for Interstitial Decongestion. JACC Basic Transl Sci. 2021 Nov 22;6(11):882-884. doi: 10.1016/j.jacbts.2021.10.003. eCollection 2021 Nov. PMID 34869952
- [Background] Aronson D. The interstitial compartment as a therapeutic target in heart failure. Front Cardiovasc Med. 2022 Aug 17;9:933384. doi: 10.3389/fcvm.2022.933384. eCollection 2022. PMID 36061549
- [Background] Mortimer PS, Rockson SG. New developments in clinical aspects of lymphatic disease. J Clin Invest. 2014 Mar;124(3):915-21. doi: 10.1172/JCI71608. Epub 2014 Mar 3. PMID 24590276
- [Background] Ratnayake CBB, Escott ABJ, Phillips ARJ, Windsor JA. The anatomy and physiology of the terminal thoracic duct and ostial valve in health and disease: potential implications for intervention. J Anat. 2018 Jul;233(1):1-14. doi: 10.1111/joa.12811. Epub 2018 Apr 10. PMID 29635686
- [Background] Witte MH, Dumont AE, Clauss RH, Rader B, Levine N, Breed ES. Lymph circulation in congestive heart failure: effect of external thoracic duct drainage. Circulation. 1969 Jun;39(6):723-33. doi: 10.1161/01.cir.39.6.723. No abstract available. PMID 5785287
- [Background] Cole WR, Witte MH, Kash SL, Rodger M, Bleisch WR, Muelheims GH. Thoracic duct-to-pulmonary vein shunt in the treatment of experimental right heart failure. Circulation. 1967 Oct;36(4):539-43. doi: 10.1161/01.cir.36.4.539. No abstract available. PMID 6041867
- [Background] Dumont AE. The flow capacity of the thoracic duct-venous junction. Am J Med Sci. 1975 May-Jun;269(3):292-301. doi: 10.1097/00000441-197505000-00001. No abstract available. PMID 1098460
- [Background] Ghelfi J, Brusset B, Teyssier Y, Sengel C, Gerster T, Girard E, Roth G, Bellier A, Bricault I, Decaens T. Endovascular Lymphatic Decompression via Thoracic Duct Stent Placement for Refractory Ascites in Patients with Cirrhosis: A Pilot Study. J Vasc Interv Radiol. 2023 Feb;34(2):212-217. doi: 10.1016/j.jvir.2022.10.030. Epub 2022 Oct 25. PMID 36306988
- [Background] Abraham WT, Jonas M, Dongaonkar RM, Geist B, Ueyama Y, Render K, Youngblood B, Muir W, Hamlin R, Del Rio CL. Direct Interstitial Decongestion in an Animal Model of Acute-on-Chronic Ischemic Heart Failure. JACC Basic Transl Sci. 2021 Nov 22;6(11):872-881. doi: 10.1016/j.jacbts.2021.09.008. eCollection 2021 Nov. PMID 34869951
- [Background] Serenyi P, Magyar Z, Szabo G. Cervical lymphato-venous shunt in treatment of ascites in caval-constricted dogs and in patients with hepatic cirrhosis. Experimental observations and 7 years clinical experience. Lymphology. 1976 Jun;9(2):53-61. PMID 957766
- [Background] Khalilzadeh O, Baerlocher MO, Shyn PB, Connolly BL, Devane AM, Morris CS, Cohen AM, Midia M, Thornton RH, Gross K, Caplin DM, Aeron G, Misra S, Patel NH, Walker TG, Martinez-Salazar G, Silberzweig JE, Nikolic B. Proposal of a New Adverse Event Classification by the Society of Interventional Radiology Standards of Practice Committee. J Vasc Interv Radiol. 2017 Oct;28(10):1432-1437.e3. doi: 10.1016/j.jvir.2017.06.019. Epub 2017 Jul 27. PMID 28757285